CLINICAL TRIAL: NCT00357838
Title: Pulse Waves and Tongue Diagnosis Differences Between Follicular and Luteal Phase in Normal Healthy Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Other Study IDs: DMR95-IRB-64
Record Dates: First submitted 2006-07-27; First posted 2006-07-28 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2006-07

CONDITIONS: Healthy
Keywords: normal healthy women

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
We hypothesized that there's difference between follicular phase and luteal phase of normal women in radial pulse waves and tongue figures.

DETAILED DESCRIPTION:
As comparing with follicular and menstrual phases of the cycle, in women during the luteal phase, the heart rate, body temperature, foot skin temperature and body weight were significantly increased. Tongue inspection and pulse examination are two methods that Chinese medical doctors are used in the diagnosis of patterns. Pulse wave analysis of the radial artery is a non-invasive, widely applicable technique for assessing cardiovascular function. Radial artery waveforms have been demonstrated being associated with the blood pressure wave of ascending and central aorta, the function of left ventricle , the arterial wall properties and the endothelial function. Even when measure locally, carries characteristic information from the whole arterial system because of reflection of waves at distinct sites of the arterial system. Examination of the changes of the arterial pulse wave between follicular phase may offer valuable insights into cardiovascular physiologic feature in menstrual cycle. The objective of this study was to test the hypothesis that the cyclic variations in hemodynamic and volume parameters during the menstrual cycle among normal healthy women. To that end we compared the following parameter of radial pulse contour between late follicular and late luteal time point: percussion wave, the difference between dicrotic wave and dicrotic notch, and the area of the wave.

ELIGIBILITY:
Inclusion Criteria:

1. Nornal period I/D=28-35/3-5 (eumenorrheic)
2. age:21-40
3. No use of oral pills in past 6 months
4. BMI1: 8.5-24.9
5. No history of smoke, alcohol or drug abuse
6. No regular exercise in past 3 month

Exclusion Criteria:

1. CVD, hepatic, renal disease
2. psychological disease
3. Thyroid disease

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Shan-Yu Su, MD, Study Chair — China Medical University Hospital
Locations (1):
- China Medical Univerity Hospital, Dawan, Taiwan

REFERENCES:
- [Background] Spaanderman ME, Van Beek E, Ekhart TH, Van Eyck J, Cheriex EC, De Leeuw PW, Peeters LL. Changes in hemodynamic parameters and volume homeostasis with the menstrual cycle among women with a history of preeclampsia. Am J Obstet Gynecol. 2000 May;182(5):1127-34. doi: 10.1067/mob.2000.105342. PMID 10819846